CLINICAL TRIAL: NCT00203957
Title: A Long-Term, Multicenter, Open-Label Safety Study With Oral 20 or 40 mg/d Doses of KW-6002 (Istradefylline) as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa Therapy
Brief Title: Study of KW-6002 (Istradefylline) in Parkinson's Disease in Patients With Motor Response Complications on Levodopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13711A; Kyowa Pharmaceuticals
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Patients who completed double-blind treatment studies 6002-US-013, 6002-US-013, 6002-US-018 immediately prior to entering this open-label trial and may have had an interuption of study drug of 14 days or less.
  Interventions: Drug: Istradefylline
- Group B (Experimental): Patients who previously completed double-blind treatment studies 6002-US-013, 6002-US-018 or 6002-EU-007 or discontinued from open label study 6002-US-007 and have had an interuption of study drug greater than 14 days.
  Interventions: Drug: Istradefylline

INTERVENTIONS:
Drug: Istradefylline — Patients will receive starting dose of 40mg/d. The allowable doses are 20 and 40mg/d
  Arms: Group A
Drug: Istradefylline — Patients will receive starting dose of 40mg/d. The allowable doses are 20 and 40mg/d
  Arms: Group B

SUMMARY:
The purpose of this study is to confirm the long term tolerability and safety of oral 20 or 40 mg/d doses of Istradefylline.

DETAILED DESCRIPTION:
This is a Phase III open-label study, in which patients with Parkinson's disease (PD) who have completed a qualifying istradefylline study will be treated with istradefylline for a period of up to one additional year. Starting dosage of istradefylline will be 40 mg/d and maintenance dosage will be at the discretion of the Investigator. The available doses for istradefylline are 20 and 40 mg/d. Open-label istradefylline treatment will be initiated after a patient has satisfied all criteria for participation.

Patients will undergo screening and baseline evaluations during which they will be assessed for eligibility. Screening procedures will vary slightly depending upon the allocation of patients to one of the following two groups:

Group A: Patients who have completed double-blind treatment studies 6002-US-0 13, 6002- US-Ol S or 6002-EU-007 immediately prior to entering this open-label trial and may have had an interruption of study drug of 14 days or less. The screening visit for these patients will correspond to the final visit of the previous istradefylline study.

Group B: Patients who have previously completed double-blind treatment studies 6002-US- 013, 6002-US-O 18 or 6002-EU-007 or discontinued from open-label study 6002-US-007 and have had an interruption of study drug greater than 14 days. Screening for these patients will occur at the Week -2 and Day -1 Visits.

Visits should occur in the ON state and procedures should be conducted in the order specified, whenever possible.

Safety outcomes will be assessed by physical examination (including neurological examination), clinical laboratory tests and 12-lead electrocardiogram (ECG) at screening and at selected subsequent scheduled visits. Vital signs, including weight, concomitant medications, and adverse events will be monitored regularly throughout the trial. Changes in anti-parkinsonian medications will be permitted at the Investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed double-blind treatment study 6002-US-0 13, 6002-US-0 18 or 6002-EU-007, or who discontinued from open-label study 6002-US-007.
* Patients who are female must be non-pregnant and non-nursing. Women of Child Bearing Potential (WOCBP) must use a reliable method of contraception (e.g., oral contraceptive or long-term injectable or implantable hormonal contraceptive, double- bather methods, such as condom and diaphragm, condom and foam, condom and sponge or intra-uterine devices) and have a negative serum (North American sites) or urine (non-North American sites) pregnancy test at screening and at baseline. Women are considered to not be of childbearing potential if they have been surgically sterilized.
* Patients who are able to give written informed consent

Exclusion Criteria:

* Group B Patients who are treated within 30 days before baseline (or five half-lives of the compound, if longer) with any investigational agent other than istradefylline
* Patients who have a history of a psychotic illness.
* Patients who are treated within three months (six months if patient was treated with depot) before baseline or during the trial with an anti-psychotic agent.
* Patients who are treated with any centrally acting drug that has known dopamine antagonist properties at therapeutic doses (e.g., buspirone, amoxapine).
* Patients who have atypical parkinsonism.
* Patients who have secondary parkinsonism variants.
* Patients who have a diagnosis of cancer or evidence of continued malignancy within five years of study enrollment (except for patients that have had basal cell carcinoma or carcinoma in situ of the cervix surgically excised).
* Patients who have a clinically significant illness of any organ system which may compromise the safety of the patient during the trial or affect the ability of the patient to complete the trial.
* Patients who, for any reason, are judged by the Investigator to be inappropriate for this trial, including a patient who is unable to communicate or to cooperate with the Investigator.
* Patients who have an ALT and/or an AST level greater than 1.5 ULN at screening will be ineligible to participate in the trial.
* Patients who have a history of drug or alcohol abuse or dependence within the last year (DSM-IVR).
* Patients with significant drug allergies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2005-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile of istradefylline | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arif Dalvi, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States